CLINICAL TRIAL: NCT02554448
Title: Detection of CTCs in Stage III Rectal Cancer Patients Undergoing Neoadjuvant Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CTC-1
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Rectal Neoplasms; Circulating Tumor Cells
Keywords: Circulating Tumor Cells; rectal Neoplasms; neoadjuvant otherapy
MeSH Terms: conditions — Rectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Circulating Tumor Cells (Experimental): Use ISET system to test the number of CTCs from patients before and during treatment.
  Interventions: Other: ISET system

INTERVENTIONS:
Other: ISET system — Use ISET system to test the number of CTCs from patients before and during treatment.

SUMMARY:
The purpose of this study is to evaluate the value of dynamic change in detecting CTCs in peripheral blood from stage III rectal cancer patients undergoing neoadjuvant Folfox treatment and chemoradiotherapy,before and after surgery.

DETAILED DESCRIPTION:
Circulating tumor cells (CTCs) have the potential to provide a surrogate for'real-time biopsy' of tumor biological activity. Enumeration of CTCs in rectal cancer patients could play an important role in diagnosis, predicting the risk for tumor recurrence and effectiveness of neoadjuvant therapy.

The investigators choose several timepoints to detect the dynamic change of CTCs,1 day before the 1st ,3rd and 5th(if the patient needs before surgery) neoadjuvant therapy course,1 day before and 7days ,3 month,6 month after surgery. Approximately 7.5-mL ethylene diamine tetraacetic acid(EDTA)-blood was drawn by vein puncture from patients with rectal cancer . Briefly, the number of CTCs will be count by the cellsearch system , recorded and analysed by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Age: >18 years old.
2. Diagnosis of stage III rectal cancer based on histology.
3. Will receive neoadjuvant treatment using Folfox or chemoradiotherapy .
4. Life expectancy: Greater than 3 months.
5. Patients have no severe inflammation, such as vasculitis.
6. Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients with other primary tumor except rectal cancer.
2. History of coagulation disorders or anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The number of Circulating Tumor Cells (CTCs) | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Yanxin Luo, PhD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliate Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
not ready to share the data